CLINICAL TRIAL: NCT02334085
Title: The Health of Women (HOW) Study
Brief Title: The Health of Women Study
Acronym: HOW
Status: Completed | Type: Observational
Sponsor: Dr. Susan Love Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 20091527
Record Dates: First submitted 2014-12-18; First posted 2015-01-08 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HOW study participants

SUMMARY:
The HOW Study is a first-of-its-kind international online study for women and men with and without a history of breast cancer. The investigators will collect information about your health, your job, your diet, and your family history, among other topics that can help us get a better understanding of breast cancer and its potential causes. Periodically, the investigators will send you questionnaires about anything and everything. All you have to do is fill them out online. It's that simple. This is a partnership and the investigators need you for the long haul. The more questionnaires you fill out, the more information the investigators will have that can help us have a better understanding of why women get breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Women
* 18 years and older

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women and men aged 18 and older, with or without breast cancer, and of all nationalities and ethnicities, from the United States and beyond, are encouraged to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 55008 (Actual)
Dates: Start 2009-08; Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Breast cancer diagnosis question | Participants will be followed for the duration of the cohort study, up to 20 years.
  In the "My Health Overview" questionnaire, the participant will be asked "have you been diagnosed with breast cancer?" Responses available are yes, no, I don't know / I can't remember, and I'd rather not say. This question will be asked in the initial questionnaire and every five years following that.

OTHER OUTCOMES:
Questions about general health status | General health status questions are available at baseline, just after enrolling in the HOW study. Participants will be followed for the duration of the cohort study, up to 20 years.
  Demographic characteristics will be obtained, questions about menstruation, pregnancy, hormone use, and lifestyle behaviors are asked in the "My Health Overview" questionnaire.
Questions about personal and family health history | Health history questions are available after the completion of the general health status questions. Participants will be followed for the duration of the cohort study, up to 20 years.
  The "My Personal and Family Health History" questionnaire asks about chronic conditions such as cancer, diabetes, hepatitis, and asthma, for the individual as well as their family members.
Questions about health, weight, and exercise | Health, weight, and exercise questions are available after the completion of the health history questions. Participants will be followed for the duration of the cohort study, up to 20 years.
  The "Health, Weight, and Exercise" questionnaire asks about sleeping patterns, weight status, a variety of exercise questions, daily activities, and prescription use.
Questions about environmental exposures | Environmental exposure questions are available after the completion of the health, weight, and exercise questions. Participants will be followed for the duration of the cohort study, up to 20 years.
  The "Environmental Exposures" questionnaire asks about cosmetic product usage, personal hygiene product usage, and second hand smoke exposure.
Questions about health symptoms (quality of life) | Health symptom questions are available at baseline, just after enrolling in the HOW study. Participants will be followed for the duration of the cohort study, up to 20 years.
  The "Quality of Life" questionnaire asks about a variety of health symptoms including problems with digestion, concentration, sex, and mental health. If you are a breast cancer survivor, you will be asked if these symptoms are related to your treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Love, MD, Principal Investigator — Dr. Susan Love Research Foundation
Locations (1):
- Dr. Susan Love Research Foundation, Santa Monica, California, United States

REFERENCES:
- See also: Related Info — https://www.healthofwomenstudy.org/